CLINICAL TRIAL: NCT05728385
Title: Impact of Modified Specific Carbohydrate Diet on Bronchial Asthma Control in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Zaki Elmeazawy, Doctor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mSCD in Asthmatic children
Record Dates: First submitted 2023-01-10; First posted 2023-02-15 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Asthma in Children
Keywords: Asthma; Children; Dietary therapy; Specific carbohydrate diet
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified SPD as adjunct to asthma medications in children (Experimental): Explore if the modified specific carbohydrate diet has an effect on asthma control in children and if it will affect the frequency, severity, and duration of asthma and thus provide it as a potential complementary treatment option for them.
  Interventions: Dietary Supplement: Modified Specific carbohydrate diet for 3 months
- Usual asthma medications only in children with moderate asthma (No Intervention): Assess control based on the usual asthma medications only

INTERVENTIONS:
Dietary Supplement: Modified Specific carbohydrate diet for 3 months — All children at the start of the study will be subjected to:
  1. Full history taking including demographic and medical history
  2. Full nutritional assessment including: Through clinical examination for any signs of vitamins and mineral deficiency, with full chest examination.
  3. Laboratory tests: Complete blood picture with differential white blood cells, and Serum IgE level
  4. At the beginning of the study and at the end
     1. The patients will be assessed using the childhood-asthma control test (C-ACT) as a subjective method
     2. Pulmonary function tests will be performed using spirometry (Spirostik, Geratherm) that includes Forced vital capacity (FVC), forced expiratory volume in the first second of FVC (FEV1), and FEV1/FVC.
     3. Anthropometric measurements: Weight, Height, and Body mass index (BMI). All measures will be plotted on specific percentile curves for age and Z score
  Arms: Modified SPD as adjunct to asthma medications in children

SUMMARY:
The aim of this study will explore if the specific carbohydrate diet has an effect on asthma control in children and if it will affect the frequency, severity, and duration of asthma and thus provide it as a potential complementary treatment option for them.

DETAILED DESCRIPTION:
This study will be carried out on 30 children with moderate persistent asthma presented to the outpatient clinic of the Pulmonology Unit, Pediatric Department, Tanta University Hospital.

All children at the start of the study will be subjected to full history taking including, full nutritional assessment, laboratory tests, Pulmonary function tests, and Anthropometric measurements

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic children with moderate persistent asthma according to the definition of National Heart, Lung, and Blood Institute guidelines, if they have daily symptoms, nighttime awakenings more than 1 time/week, but not nightly, daily use of short-acting beta-agonist for symptom control, some limitations of normal activities, and Forced Expiratory Volume in 1 second (FEV1)60-80%.
* Children aged from 6 to 18 years.
* The children are included only if parents and children are strongly motivated to try a dietary intervention (mSCD) as a complementary treatment.

Exclusion Criteria:

* Children with chronic lung disease, immunodeficiency, major thoracic deformities, neuromuscular, cardiovascular, digestive, rheumatic, osteoarticular, or genetic syndromes or any adverse health conditions that can affect nutritional status were excluded from the study.
* Children excluded if parents and children are not motivated to try a dietary intervention (mSCD) as a complementary treatment or who failed to have regular outpatient follow-up visits.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Childhood-asthma control test (C-ACT) as a subjective method | Baseline (three months)
  The C-ACT consists of a 7-item validated questionnaire, addresses the previous 4 weeks and is divided into two parts. One part is filled in by the child and consists of four questions on perception of asthma control, limitation of activities, coughing and awakenings at night. Each question has four response options. The second part is filled in by the parent or caregiver and consists of three questions (daytime complaints, daytime wheezing and awakenings at night) with six response options. The sum of all scores yields the C-ACT score, ranging from 0 (poorest asthma control) to 27 (optimal asthma control). A cut-off point ≤ 19indicates uncontrolled asthma

SECONDARY OUTCOMES:
FEV1 | three months
  Will be performed using spirometry (Spirostik, Geratherm) to measure forced expiratory volume at the end of the first second.
FVC | three months
  Will be performed using spirometry (Spirostik, Geratherm) to measure forced vital capacity.
FEV1/FVC ratio | three months
  Will be performed using spirometry (Spirostik, Geratherm) to measure the ratio of forced expiratory volume at the end of first second to the forced vital capacity.

REFERENCES:
- [Background] Reddel HK, Bacharier LB, Bateman ED, Brightling CE, Brusselle GG, Buhl R, Cruz AA, Duijts L, Drazen JM, FitzGerald JM, Fleming LJ, Inoue H, Ko FW, Krishnan JA, Levy ML, Lin J, Mortimer K, Pitrez PM, Sheikh A, Yorgancioglu AA, Boulet LP. Global Initiative for Asthma Strategy 2021: Executive Summary and Rationale for Key Changes. J Allergy Clin Immunol Pract. 2022 Jan;10(1S):S1-S18. doi: 10.1016/j.jaip.2021.10.001. Epub 2021 Oct 28. PMID 34718211
- [Background] Bedard A, Li Z, Ait-Hadad W, Camargo CA Jr, Leynaert B, Pison C, Dumas O, Varraso R. The Role of Nutritional Factors in Asthma: Challenges and Opportunities for Epidemiological Research. Int J Environ Res Public Health. 2021 Mar 15;18(6):3013. doi: 10.3390/ijerph18063013. PMID 33804200
- [Background] Beasley R, Semprini A, Mitchell EA. Risk factors for asthma: is prevention possible? Lancet. 2015 Sep 12;386(9998):1075-85. doi: 10.1016/S0140-6736(15)00156-7. PMID 26382999
- [Background] Julia V, Macia L, Dombrowicz D. The impact of diet on asthma and allergic diseases. Nat Rev Immunol. 2015 May;15(5):308-22. doi: 10.1038/nri3830. PMID 25907459
- [Background] Guilleminault L, Williams EJ, Scott HA, Berthon BS, Jensen M, Wood LG. Diet and Asthma: Is It Time to Adapt Our Message? Nutrients. 2017 Nov 8;9(11):1227. doi: 10.3390/nu9111227. PMID 29117118
- [Background] Loverdos K, Bellos G, Kokolatou L, Vasileiadis I, Giamarellos E, Pecchiari M, Koulouris N, Koutsoukou A, Rovina N. Lung Microbiome in Asthma: Current Perspectives. J Clin Med. 2019 Nov 14;8(11):1967. doi: 10.3390/jcm8111967. PMID 31739446
- [Background] Wahbeh GT, Ward BT, Lee DY, Giefer MJ, Suskind DL. Lack of Mucosal Healing From Modified Specific Carbohydrate Diet in Pediatric Patients With Crohn Disease. J Pediatr Gastroenterol Nutr. 2017 Sep;65(3):289-292. doi: 10.1097/MPG.0000000000001619. PMID 28825776
- [Background] Suskind DL, Lee D, Kim YM, Wahbeh G, Singh N, Braly K, Nuding M, Nicora CD, Purvine SO, Lipton MS, Jansson JK, Nelson WC. The Specific Carbohydrate Diet and Diet Modification as Induction Therapy for Pediatric Crohn's Disease: A Randomized Diet Controlled Trial. Nutrients. 2020 Dec 6;12(12):3749. doi: 10.3390/nu12123749. PMID 33291229
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040